CLINICAL TRIAL: NCT01485068
Title: Assessment of the Safety and Efficacy of the Danubio Paclitaxel-Eluting Balloon for the Treatment of In-Stent Restenosis Lesions in Native Coronary Arteries.
Brief Title: Safety and Efficacy Study of the DANUBIO Paclitaxel Eluting Balloon in In-Stent Restenosis Lesions (DEBREST)
Acronym: DEBREST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MINVASYS (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIN1102
Record Dates: First submitted 2011-11-14; First posted 2011-12-05 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2013-11

CONDITIONS: In-stent Coronary Artery Restenosis
Keywords: Restenosis; Paclitaxel-eluting balloon; Angioplasty; Coronary artery disease; Coronary artery stenosis
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Danubio (Experimental)
  Interventions: Device: Danubio paclitaxel-eluting balloon

INTERVENTIONS:
Device: Danubio paclitaxel-eluting balloon — Inflation of the Danubio Paclitaxel Eluting Balloon in in-stent restenosis lesions.

SUMMARY:
The purpose of this study is to assess safety and efficacy of the Danubio Paclitaxel Eluting Balloon for the treatment of In-Stent Restenosis lesions in native coronary arteries.

DETAILED DESCRIPTION:
The DEBREST clinical trial is a prospective, non-randomized, multicenter, interventional study evaluating the investigational Danubio Paclitaxel Eluting Coronary Balloon in patients with in-stent restenosis (ISR) lesion(s) with reference vessel diameter ≥2.5 mm and ≤3.5 mm. The trial will allow the treatment of up to two ISR (either Bare Metal Stent (BMS) or Drug Eluting Stent (DES) ISR) per patient in native coronary arteries with mandatory predilatation with a conventional balloon.

The DEBREST clinical trial will enroll 60 patients. All patients will receive Quantitative Coronary Angiography (QCA) before and after Drug-Eluting Balloon (DEB) inflation and at 6 months follow-up. All patients will have a clinical follow-up at 1, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Restenotic lesion in a native coronary artery.
2. First ISR after BMS or DES implantation.
3. Reference diameter > 2.5 and ≤ 3.5mm.
4. Target lesion length: ≤ 21mm.
5. Up to three restenotic lesions per patient.
6. Single restenotic lesion per vessel.
7. The lesion must be treated with the trial device Danubio.
8. During the index procedure, in case of

   1. Treatment of a lesion in a vessel other than the target vessel or,
   2. Treatment of a lesion in the target vessel proximal or distal to the target restenotic lesion, The treatment of the non-target lesion must be successfully performed with a Drug-Eluting Stent before the treatment of the target lesion (residual stenosis <30%; stent well deployed; no residual dissection; normal TIMI flow; no chest pain; ECG unchanged compared to pre-procedural ECG).
9. Successful predilatation with a conventional balloon providing good angiographic result (i.e. absence of dissection, TIMI > III).
10. The patient is at least 18 years of age.
11. Non menopausal women must provide a negative pregnancy test and use a double contraception until the end of the study.
12. The patient has clinical evidence of ischemic heart disease, stable or unstable angina with signs of ischemia, silent ischemia, or a positive functional test.
13. The patient is an acceptable candidate for percutaneous transluminal coronary angioplasty (PTCA), stenting, and emergent coronary artery bypass graft (CABG) surgery.
14. The patient or patient's legal representative has been informed of the nature of the trial and agrees to its provisions and has provided written informed consent as approved by the Ethics Committee (EC).
15. The patient agrees to return to the same research facility for required angiographic post-procedure follow-up visit at 6 months .

Exclusion Criteria:

1. Bifurcation lesion(s) including left main.
2. The Danubio covers beyond the lesion proximally and distally with < 2 mm.
3. Heavily calcified lesions.
4. Severe tortuous lesions.
5. Evidence of extensive thrombosis or dissection within target vessel before the intervention.
6. Documented Left Ventricular Ejection Fraction (LVEF) < 30% at most recent evaluation.
7. A known hypersensitivity or contraindication to aspirin, heparin or bivaluridin, ticlopidine or clopidogrel, paclitaxel or drugs in similar class, contrast media, which cannot be adequately pre-medicated.
8. Chronic total occlusion (CTO).
9. A serum creatinine level > 2.0 mg/dL within seven days prior to index procedure.
10. Evidence of an acute MI within 72 hours of the intended index procedure (according to ARC definition).
11. Planned PCI of any vessel within 30 days post-procedure.
12. Surgery 30 days prior to this PCI or anticipated surgery 6-months post this PCI.
13. During the index procedure, the target lesion requires treatment with a device other than PTCA prior to use of Danubio (including but not limited to cutting balloon, any atherectomy, any laser, thrombectomy, etc.).
14. Second restenotic lesion requiring treatment in target vessel.
15. History of a stroke or transient ischemic attack (TIA) within the prior 6 months
16. Active peptic ulcer or upper gastrointestinal (GI) bleeding within the prior 6 months.
17. History of bleeding diathesis or coagulopathy or will refuse blood transfusions.
18. Concurrent medical condition with a life expectancy of less than 12 months.
19. Any previous or planned treatment of the target vessel with anti-restenotic therapies including, but not limited to brachytherapy.
20. Currently participating in an investigational drug or another device trial that has not completed the primary endpoint or that clinically interferes with the current trial endpoints; or requires coronary angiography, IVUS or other coronary artery imaging procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-03; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
In-stent Late Lumen Loss (mm) | 6 months post-procedure (up to 26 weeks)
  In-stent Late Lumen Loss by Quantitative Coronary Angiography (QCA)

SECONDARY OUTCOMES:
In-segment Late Lumen Loss (mm) | 6 months post-procedure (up to 26 weeks)
  In-segment Late Lumen Loss by QCA.
Angiographic binary restenosis rate (%) | 6 months post-procedure (up to 26 weeks)
  Angiographic binary restenosis rate (%) by QCA.
Major Adverse Cardiac Event (MACE) rate | In-hospital, 1, 6 and 12 months post-procedure.
  MACE defined as death, Myocardial Infarction (MI, Q waves and non-Q waves), emergent cardiac bypass surgery, or any target lesion revascularization (repeat Percutaneous transluminal coronary angioplasty (PTCA) or Coronary artery bypass grafting (CABG)).
Clinically-driven Target Lesion Revascularization (TLR) | 1, 6 and 12 months post-procedure
Target Vessel Failure (TVF) | 1, 6 and 12 months post-procedure
Target Vessel Revascularization (TVR) | 1, 6 and 12 months post-procedure
Angiographic success | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Jacques BERLAND, MD, Principal Investigator — Clinique Saint Hilaire - ROUEN
Locations (8):
- France (8):
  - Hôpital Privé d'Antony, Antony
  - Centre Hospitalier privé Saint-Martin, Caen
  - Centre cardiologique d'Evecquemont, Évecquemont
  - Centre Hospitalier d'Haguenau, Haguenau
  - Les Franciscaines, Nîmes
  - Polyclinique les Fleurs, Ollioules
  - Clinique Saint-Pierre, Perpignan
  - Clinique Saint-Martin, Pessac